CLINICAL TRIAL: NCT03400319
Title: Obstructive Sleep Apnoea in Adolescents With Thoracic Aortic Aneurysm
Acronym: OSA in TAA
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0035 CTRL
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Thoracic Aortic Aneurysm Without Rupture; Obstructive Sleep Apnea
Keywords: Thoracic Aortic Aneurysm; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracic Aortic Aneurysm: Patients with Thoracic Aortic Aneurysm: Women: at the level of the sinus of valsalva ≥39mm, or ascending aorta ≥42mm. Men: at the level of the sinus of valsalva ≥44mm, or ascending aorta ≥46mm.
- No Thoracic Aortic Aneurysm: Patients without Thoracic Aortic Aneurysm: Women: at the level of the sinus of valsalva <39mm, or ascending aorta <42mm. Men: at the level of the sinus of valsalva <44mm, or ascending aorta <46mm.

SUMMARY:
The objective of this prospective cohort study is to determine the prevalence of obstructive sleep apnoea (OSA) in patients with and without thoracic aortic aneurysm.

DETAILED DESCRIPTION:
The objective of this prospective cohort study is to determine the prevalence of obstructive sleep apnoea (OSA) in patients with and without thoracic aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Diagnosis of thoracic aortic aneurysm defined by the following parameters:

Women: at the level of the sinus of valsalva ≥39mm, or ascending aorta ≥42mm. (for controls: <39mm and <42mm respectively); Men: at the level of the sinus of valsalva ≥44mm, or ascending aorta ≥46mm. (for controls: <44mm and <46mm respectively)

Exclusion Criteria:

* Patients on continuous positive airway pressure (CPAP) therapy for OSA at baseline.
* Patients with known central sleep apnoea.
* Patients on morphine or other opioid medication, heroin addiction, alcohol addiction.
* Patients with moderate or severe aortic regurgitation.
* Patients with moderate or severe aortic stenosis.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without Thoracic Aortic Aneurysm
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2014-07-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Obstructive Sleep Apnea | Baseline
  Prevalence of Obstructive Sleep Apnea according to a Sleep study (The ApneaLink™)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No